CLINICAL TRIAL: NCT07013552
Title: Oritavancin as a Therapeutic Regimen for Cardiac Implantable Electronic Devices Infections With Multidrug-resistant Gram-positive Cocci
Brief Title: Oritavancin for CIED Infections With MDR Gram-positive Cocci
Acronym: ORI-4-CIEDi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPOD.07.07-IW.07-0004/24
Record Dates: First submitted 2025-05-12; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Implantable Electronic Device Infections; Infective Endocarditis; Multidrug-resistant Bacteria Screening; Gram Positive Bacterial Infection; Antibiotic Resistant Strain; Antibiotic Therapy; Healthcare Associated Infections
Keywords: Cardiac implantable electronic device; Gram-positive cocci; Health-care associated infections; Lead-related infective endocarditis; Multidrug-resistant bacteria; Pocket infection
MeSH Terms: conditions — Endocarditis; Gram-Positive Bacterial Infections; Cross Infection

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to the intervention and control groups.
  Experimental group:
  Oritavancin dosage in superficial ABSSSI or PI: Single dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion.
  Oritavancin dosage in LRIE: First dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion, subsequent doses of 800 mg (2 vials) administered as a 2-3 hour intravenous infusion at 7-day intervals, to achieve the required duration of drug therapy of 2-6 weeks (counted from the day of transvenous lead extraction).
  Control group:
  Vancomycin dosage: Repeated doses of 15-20 mg/kg body weight every 8-12 hours administered as an hourly intravenous infusion for 7-10 days in ABSSSI, for 10-14 days in PI, and for 2-6 weeks in LRIE.
Masking Description: The study will be blinded only at the randomization stage. A different time model for antibiotic dosing does not allow for blinding of the Care Provider and allows the Participant to easily identify the type of antibiotic administered based on the information obtained in the consent form for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with a long half-life antibiotic - oritavancin (Tenkasi) (Experimental): Patients with CIED infection with MDR Gram-positive cocci treated with a long half-life lipoglycopeptide antibiotic - oritavancin
  Interventions: Drug: Administration of a single or repeated dose of a long half-life antibiotic - oritavancin
- Patients treated with a short half-life antibiotic - vancomycin (Vancomycin) (Active Comparator): Patients with CIED infection with MDR Gram-positive cocci treated with a short half-life glycopeptide antibiotic - vancomycin
  Interventions: Drug: Administration of a repeated dose of a short half-life antibiotic - vancomycin

INTERVENTIONS:
Drug: Administration of a single or repeated dose of a long half-life antibiotic - oritavancin — Intravenous administration of a single or repeated dose of lipoglycopeptide antibiotic - oritavancin.
  In superficial ABSSSI or PI: Single dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion in 5% glucose solution.
  In LRIE: First dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion in 5% glucose solution, subsequent doses of 800 mg (2 vials) administered as a 2-3 hour intravenous infusion at 7-day intervals, to achieve the required duration of drug therapy of 2-6 weeks (counted from the day of transvenous lead extraction).
  Arms: Patients treated with a long half-life antibiotic - oritavancin (Tenkasi)
Drug: Administration of a repeated dose of a short half-life antibiotic - vancomycin — Intravenous administration of repeated doses of glycopeptide antibiotic - vancomycin.
  Repeated doses of 15-20 mg/kg body weight every 8-12 hours administered as an hourly intravenous infusion in 0.9% sodium chloride solution, under monitoring the drug concentration in serum, for 7-10 days in ABSSSI, for 10-14 days in PI, and for 2-6 weeks in LRIE (counted from the day of transvenous lead extraction).
  Arms: Patients treated with a short half-life antibiotic - vancomycin (Vancomycin)

SUMMARY:
The study aimed to conduct a randomized, non-inferiority controlled trial to compare the short- and medium-term efficacy and safety of two antibiotic dosage regimens in cardiac implantable electronic devices (CIED) infections with multidrug-resistant Gram-positive cocci: 1) single-dose therapy with a long-half-life antibiotic (oritavancin) vs. standard 7-14 days of therapy with a short-half-life antibiotic (vancomycin) for CIED surgical incision site or pocket infection; and 2) fractionated therapy with a long-half-life antibiotic (oritavancin) at seven-day intervals compared to standard therapy with a short-half-life antibiotic (vancomycin) fractionated in 2-3 daily doses in cases of lead-related infectious endocarditis.

DETAILED DESCRIPTION:
Study Objectives:

This study's purpose is to evaluate the safety and efficacy of two antibiotic dosage regimens in a pilot study of cardiac implantable electronic devices (CIED) infections with multidrug-resistant (MDR) Gram-positive cocci.

Study Design:

This study is a single-center randomized, non-inferiority, control trial comparing the efficacy and safety of two antibiotic dosage regimens with a long-half-life antibiotic (oritavancin, experimental group) vs. standard therapy with a short-half-life antibiotic (vancomycin, control group).

Study Assumptions:

The investigators assumed that the efficacy of oritavancin therapy administered as a single intravenous infusion (for surgical incision site infection or pocket infection) or in fractionated doses administered at seven-day intervals (for lead-related infectious endocarditis) would be non-inferior to the efficacy of standard vancomycin therapy administered daily at 8-12 hour intervals and that there would be no difference in the safety profile between the two therapies.

Patient Population:

Patients aged ≥18 with CIED surgical incision site infection (i.e., superficial acute bacterial skin and skin structure infections, ABSSSI) or deep infections of the generator pocket (PI) complicated or not with lead-related infectious endocarditis (LRIE) (optional) with multidrug-resistant (MDR) Gram-positive cocci.

The planned size of the group in the pilot study is 50-100. The planned recruitment period is 15 months, and the observation period is 3 months.

Once all inclusion criteria and none of the exclusion criteria are met, patients who have given written informed consent to participate in the study will be randomly assigned to the experimental group and the control group to achieve a 1:1 group size ratio.

Intervention:

The diagnostic and surgical approach and the duration of antibiotic treatment will be determined depending on the etiological factor and clinical indications by the consensus of European Heart Rhythm Association and Heart Rhythm Society experts on cardiovascular implantable electronic device lead management and extraction and the European Society of Cardiology guidelines for the treatment of infective endocarditis.

The intervention under investigation (experimental) will be administering a single or repeated dose of oritavancin.

The standard intervention will be administering of repeated doses of vancomycin.

Experimental group - Oritavancin dosage:

1. in superficial ABSSSI: Single dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion in 5% glucose solution (infusion volume: 1,000 ml);
2. in isolated PI: Single dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion in 5% glucose solution (infusion volume: 1,000 ml);
3. in LRIE: First dose of 1,200 mg (3 vials) administered as a 3-hour intravenous infusion in 5% glucose solution (infusion volume: 1,000 ml), subsequent doses of 800 mg (2 vials) administered as a 2-3 hour intravenous infusion at 7-day intervals, to achieve the required duration of drug therapy of 2-6 weeks (counted from the day of TLE).

Control group - Vancomycin dosage:

1. in superficial ABSSSI: Repeated doses of 15-20 mg/kg body weight every 8-12 hours (maximum 3,000 mg/day for patients with normal renal function) administered as an hourly intravenous infusion in 0.9% sodium chloride solution (infusion volume: 500-1,000 ml), under monitoring the drug concentration in serum, for 7-10 days (calculated from the beginning of antibiotic therapy, not less than seven days from surgical tissue debridement, if required);
2. in isolated PI: Repeated doses of 15-20 mg/kg body weight every 8-12 hours (maximum 3,000 mg/day for patients with normal renal function) administered as an hourly intravenous infusion in 0.9% sodium chloride solution (infusion volume: 500-1,000 ml), under monitoring the drug concentration in serum, for 10-14 days (counted from the day of surgical debridement of the generator pocket and TLE, if possible);
3. in LRIE: Repeated doses of 15-20 mg/kg body weight every 8-12 hours (maximum 3,000 mg/day for patients with normal renal function) administered as an hourly intravenous infusion in 0.9% sodium chloride solution (infusion volume: 500-1,000 ml), under monitoring the drug concentration in serum, to achieve the required pharmacotherapy time of 2-6 weeks (counted from the day of surgical debridement of the incision site and TLE).

Observation:

Observation will include

1. Physical examination with the assessment of the CIED implantation site;
2. Routine laboratory tests, including blood count, C-reactive protein (mg/l), procalcitonin (ng/ml), plasma creatinine (mg/dl);
3. Transthoracic echocardiogram with the assessment of bacterial vegetations;
4. Transesophageal echocardiogram with the assessment of bacterial vegetations, with particular emphasis on the tricuspid valve and CIED leads;
5. PET/CT examination with 18F-FDG or SPECT/CT using radioisotope-labeled leukocytes (depending on clinical indications).

Evaluation will be performed at 72-120 hours of therapy, after 5-7 and 14 days of therapy, and after 1 and 3 months of therapy, with endpoints assessed at 3 months.

Primary endpoints will include a complete cure rate and serious treatment-related adverse events at 3 months of follow-up.

Secondary endpoints will include clinical response rates, worsening or recurrence of infection despite drug therapy (including those resulting in rehospitalization and requiring alternative antibiotic therapy), and time to clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Completed 18 years of age
2. Presence of signs and symptoms of superficial ABSSSI or PI in the form of a) redness/warmth/swelling/pain or b) separation of the edges of the surgical incision with signs of inflammation or the need for repeated surgical debridement of the wound or c) the presence of decubitus of the skin and subcutaneous tissue in area of the generator or skin abscess/erosion of the device pocket, with purulent discharge from the wound or discharge giving a positive microbial culture
3. Probable/ definite diagnosis of right-sided LRIE according to modified Dukes criteria (optional criterion)
4. Suspected/confirmed infection with drug-resistant Gram-positive cocci, i.e., Staphylococcus spp. (Stahphylococcus aureus or coagulase-negative staphylococci), Streptococcus spp. or Enterococcus spp. sensitive to oritavancin
5. Suspected/confirmed infection with Gram-positive cocci, i.e., Staphylococcus spp., Streptococcus spp., Enterococcus spp., sensitive to vancomycin or oritavancin and beta-lactam antibiotics in patients with a history of type I anaphylaxis to penicillin.

Exclusion Criteria:

1. Suspected/confirmed infection with Gram-positive or Gram-negative bacilli or anaerobic bacteria
2. Suspected/confirmed community-acquired infection or infection with Gram-positive cocci sensitive to betalactam antibiotics, including penicillin, ampicillin, or methicillin, based on empirical data or cultures (does not apply to patients with a history of type I anaphylaxis to penicillin)
3. Confirmed resistance of Gram-positive cocci, which are the etiological factor of the infection, to vancomycin and oritavancin.
4. History of hypersensitivity to oritavancin or another lipoglycopeptide antibiotic (applies to the experimental group only)
5. History of hypersensitivity to vancomycin or another glycopeptide antibiotics (applies to the control group only)
6. No possibility of temporarily interrupting/initiating alternative therapy to intravenous infusion of unfractionated heparin
7. Pregnancy or breastfeeding
8. Lack of informed written consent of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Co-primary efficacy endpoint - treatment success rate | 3 months
  Treatment success will be defined as obtaining a clinical response and no recurrence of infection at the same site or the site of CIED reimplantation within three months of F/U.
Co-primary safety endpoint - no treatment-related Serious Adverse Events | 3 months
  Any adverse event classified as grade 3-5 according Health Technology Assessment report developed by the Agency for Health Technology Assessment and Tariff System (Poland) and related to using the investigational product (scores of 3-5) will be counted as a safety endpoint.

SECONDARY OUTCOMES:
Clinical response rate | 3 months
  Clinical response will be defined as follows:
  1. In the case of ABSSSI: a reduction in the size of the inflammatory lesion by at least 20% compared to the baseline after 48-72 hours of antibiotic therapy (in the case of conservative treatment) or the resolution of ABSSSI/complete healing of the surgical wound assessed after 7-10 days.
  2. In the case of isolated PI: a resolution of fever and reduction of inflammatory parameters by ≥50% after 72-120 hours of antibiotic therapy and complete healing of the surgical wound assessed after 10-14 days.
  3. In the case of PI complicated by LRIE: a reduction of inflammatory parameters by ≥50% after 72-120 hours of antibiotic therapy, negative control blood cultures after 72 hours, and resolution of fever by the 7th day, complete healing of the surgical wound after 10-14 days and resolution and absence of new echocardiographic signs of infection after the end of antibiotic therapy.
Median time to clinical response | 3 months
  Median time to clinical response defined as above and given in hours or days (as required).
Recurrent infection rate | 3 months
  Recurrence of infection will be defined as CIED infection occurring within three months of the completion of previous treatment, caused by the persistence of bacteria with the same phenotype in the skin and subcutaneous tissue, the device pocket, intracardiac leads, the right-sided endocardium or tricuspid valve.
Rehospitalization rate due to recurrent infection | 3 months
  Hospitalization due to recurrent infection will be defined as a hospital stay resulting from the need for repeated antibiotic administration or repeated surgical intervention related to recurrent infection in the form of ABSSSI, PI, or LRIE (as outlined in point 5).
Proportion of cases in which infection worsened from superficial or local to systemic despite drug therapy | 3 months
  A case in which an infection escalates from superficial or localized to systemic despite receiving drug therapy will be defined as a situation in which, after performing all planned initial tests, including transesophageal echocardiography and blood cultures, ABSSSI or PI will be diagnosed. However, during further follow-up, new clinical symptoms, laboratory tests, or imaging studies will indicate the development of LRIE.
Proportion of cases in which alternative "rescue" antibiotic therapy was used due to treatment failure | 3 months
  Treatment failure was defined as a lack of clinical response or worsening of infection despite adequate antibiotic therapy and surgical treatment (if necessary) or the need for alternative "rescue" antibiotic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Sarecka-Hujar, Professor, Principal Investigator — Department of Basic Biomedical Science, Faculty of Pharmaceutical Sciences in Sosnowiec, Medical University of Silesia, Poland
Locations (1):
- Department of Electrocardiology and Heart Failure, Medical University of Silesia in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The raw IPD data that underlie results in a publications will be openly available.
Supporting Information: Study Protocol
Time Frame: A link to the IPD data that underlie results in a publication will be available immediately after the manuscript is accepted and published.
Access Criteria: The raw IPD data and supporting Information will be openly available in the Polish Platform of Medical Research (https://ppm.edu.pl/search/researchdata?ps=20&t=simple&showRel=false&lang=pl&qp=&cid=1577414) under the CC BY license.

REFERENCES:
- [Background] Gladysz-Wanha S, Joniec M, Wanha W, Pilat E, Drzewiecka A, Gardas R, Biernat J, Weglarzy A, Golba KS. Transvenous lead extraction safety and efficacy in infected and noninfected patients using mechanical-only tools: Prospective registry from a high-volume center. Heart Rhythm. 2024 Apr;21(4):427-435. doi: 10.1016/j.hrthm.2023.12.015. Epub 2023 Dec 28. PMID 38157921
- [Background] Olsen T, Jorgensen OD, Nielsen JC, Thogersen AM, Philbert BT, Johansen JB. Incidence of device-related infection in 97 750 patients: clinical data from the complete Danish device-cohort (1982-2018). Eur Heart J. 2019 Jun 14;40(23):1862-1869. doi: 10.1093/eurheartj/ehz316. PMID 31155647
- [Background] Stewart CL, Turner MS, Frens JJ, Snider CB, Smith JR. Real-World Experience with Oritavancin Therapy in Invasive Gram-Positive Infections. Infect Dis Ther. 2017 Jun;6(2):277-289. doi: 10.1007/s40121-017-0156-z. Epub 2017 Apr 6. PMID 28386776
- [Background] Morrisette T, Miller MA, Montague BT, Barber GR, McQueen RB, Krsak M. On- and off-label utilization of dalbavancin and oritavancin for Gram-positive infections. J Antimicrob Chemother. 2019 Aug 1;74(8):2405-2416. doi: 10.1093/jac/dkz162. PMID 31322694
- [Background] Rubino CM, Bhavnani SM, Moeck G, Bellibas SE, Ambrose PG. Population pharmacokinetic analysis for a single 1,200-milligram dose of oritavancin using data from two pivotal phase 3 clinical trials. Antimicrob Agents Chemother. 2015;59(6):3365-72. doi: 10.1128/AAC.00176-15. Epub 2015 Mar 30. PMID 25824211
- [Background] Carvalhaes CG, Sader HS, Streit JM, Castanheira M, Mendes RE. Activity of Oritavancin against Gram-Positive Pathogens Causing Bloodstream Infections in the United States over 10 Years: Focus on Drug-Resistant Enterococcal Subsets (2010-2019). Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0166721. doi: 10.1128/AAC.01667-21. Epub 2021 Nov 22. PMID 34807761
- [Background] Tacconelli E, Carrara E, Savoldi A, Harbarth S, Mendelson M, Monnet DL, Pulcini C, Kahlmeter G, Kluytmans J, Carmeli Y, Ouellette M, Outterson K, Patel J, Cavaleri M, Cox EM, Houchens CR, Grayson ML, Hansen P, Singh N, Theuretzbacher U, Magrini N; WHO Pathogens Priority List Working Group. Discovery, research, and development of new antibiotics: the WHO priority list of antibiotic-resistant bacteria and tuberculosis. Lancet Infect Dis. 2018 Mar;18(3):318-327. doi: 10.1016/S1473-3099(17)30753-3. Epub 2017 Dec 21. PMID 29276051
- [Background] Lupia T, De Benedetto I, Bosio R, Shbaklo N, De Rosa FG, Corcione S. Role of Oritavancin in the Treatment of Infective Endocarditis, Catheter- or Device-Related Infections, Bloodstream Infections, and Bone and Prosthetic Joint Infections in Humans: Narrative Review and Possible Developments. Life (Basel). 2023 Apr 6;13(4):959. doi: 10.3390/life13040959. PMID 37109488
- [Background] Thomas G, Henao-Martinez AF, Franco-Paredes C, Chastain DB. Treatment of osteoarticular, cardiovascular, intravascular-catheter-related and other complicated infections with dalbavancin and oritavancin: A systematic review. Int J Antimicrob Agents. 2020 Sep;56(3):106069. doi: 10.1016/j.ijantimicag.2020.106069. Epub 2020 Jun 27. PMID 32603683
- [Background] Esposito S, Blasi F, Curtis N, Kaplan S, Lazzarotto T, Meschiari M, Mussini C, Peghin M, Rodrigo C, Vena A, Principi N, Bassetti M. New Antibiotics for Staphylococcus aureus Infection: An Update from the World Association of Infectious Diseases and Immunological Disorders (WAidid) and the Italian Society of Anti-Infective Therapy (SITA). Antibiotics (Basel). 2023 Apr 12;12(4):742. doi: 10.3390/antibiotics12040742. PMID 37107104
- [Background] Corey GR, Arhin FF, Wikler MA, Sahm DF, Kreiswirth BN, Mediavilla JR, Good S, Fiset C, Jiang H, Moeck G, Kabler H, Green S, O'Riordan W; SOLO I, SOLO II Investigators. Pooled analysis of single-dose oritavancin in the treatment of acute bacterial skin and skin-structure infections caused by Gram-positive pathogens, including a large patient subset with methicillin-resistant Staphylococcus aureus. Int J Antimicrob Agents. 2016 Nov;48(5):528-534. doi: 10.1016/j.ijantimicag.2016.07.019. Epub 2016 Sep 13. PMID 27665522
- [Background] Giske CG, Turnidge J, Canton R, Kahlmeter G; EUCAST Steering Committee. Update from the European Committee on Antimicrobial Susceptibility Testing (EUCAST). J Clin Microbiol. 2022 Mar 16;60(3):e0027621. doi: 10.1128/JCM.00276-21. Epub 2021 Aug 4. PMID 34346716
- [Background] Delgado V, Ajmone Marsan N, de Waha S, Bonaros N, Brida M, Burri H, Caselli S, Doenst T, Ederhy S, Erba PA, Foldager D, Fosbol EL, Kovac J, Mestres CA, Miller OI, Miro JM, Pazdernik M, Pizzi MN, Quintana E, Rasmussen TB, Ristic AD, Rodes-Cabau J, Sionis A, Zuhlke LJ, Borger MA; ESC Scientific Document Group. 2023 ESC Guidelines for the management of endocarditis. Eur Heart J. 2023 Oct 14;44(39):3948-4042. doi: 10.1093/eurheartj/ehad193. No abstract available. PMID 37622656
- [Background] Milman A, Wieder-Finesod A, Zahavi G, Meitus A, Kariv S, Shafir Y, Beinart R, Rahav G, Nof E. Complicated Pocket Infection in Patients Undergoing Lead Extraction: Characteristics and Outcomes. J Clin Med. 2023 Jun 29;12(13):4397. doi: 10.3390/jcm12134397. PMID 37445433
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379
- [Background] Blomstrom-Lundqvist C, Traykov V, Erba PA, Burri H, Nielsen JC, Bongiorni MG, Poole J, Boriani G, Costa R, Deharo JC, Epstein LM, Saghy L, Snygg-Martin U, Starck C, Tascini C, Strathmore N; ESC Scientific Document Group. European Heart Rhythm Association (EHRA) international consensus document on how to prevent, diagnose, and treat cardiac implantable electronic device infections-endorsed by the Heart Rhythm Society (HRS), the Asia Pacific Heart Rhythm Society (APHRS), the Latin American Heart Rhythm Society (LAHRS), International Society for Cardiovascular Infectious Diseases (ISCVID) and the European Society of Clinical Microbiology and Infectious Diseases (ESCMID) in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). Europace. 2020 Apr 1;22(4):515-549. doi: 10.1093/europace/euz246. PMID 31702000
- [Background] Polewczyk A, Jachec W, Polewczyk M, Nowosielecka D, Brzozowski W, Kutarski A. Outcomes in patients with definite and possible infective endocarditis related to a cardiac implantable electronic device. Pol Arch Intern Med. 2024 Aug 8;134(7-8):16775. doi: 10.20452/pamw.16775. Epub 2024 Jun 17. PMID 38895973
- [Background] Bongiorni MG, Kennergren C, Butter C, Deharo JC, Kutarski A, Rinaldi CA, Romano SL, Maggioni AP, Andarala M, Auricchio A, Kuck KH, Blomstrom-Lundqvist C; ELECTRa Investigators. The European Lead Extraction ConTRolled (ELECTRa) study: a European Heart Rhythm Association (EHRA) Registry of Transvenous Lead Extraction Outcomes. Eur Heart J. 2017 Oct 21;38(40):2995-3005. doi: 10.1093/eurheartj/ehx080. PMID 28369414
- [Background] Chmielarczyk A, Pomorska-Wesolowska M, Romaniszyn D, Wojkowska-Mach J. Healthcare-Associated Laboratory-Confirmed Bloodstream Infections-Species Diversity and Resistance Mechanisms, a Four-Year Retrospective Laboratory-Based Study in the South of Poland. Int J Environ Res Public Health. 2021 Mar 9;18(5):2785. doi: 10.3390/ijerph18052785. PMID 33803428
- [Background] Joshi S, Shallal A, Zervos M. Vancomycin-Resistant Enterococci: Epidemiology, Infection Prevention, and Control. Infect Dis Clin North Am. 2021 Dec;35(4):953-968. doi: 10.1016/j.idc.2021.07.002. PMID 34752227
- [Background] Cerini P, Meduri FR, Tomassetti F, Polidori I, Brugneti M, Nicolai E, Bernardini S, Pieri M, Broccolo F. Trends in Antibiotic Resistance of Nosocomial and Community-Acquired Infections in Italy. Antibiotics (Basel). 2023 Mar 24;12(4):651. doi: 10.3390/antibiotics12040651. PMID 37107013
- See also: Lekooporność Streptococcus pneumoniae: częstość występowania, mechanizmy, znaczenie kliniczne. Aktualności Narodowego Programu Ochrony Antybiotyków 2019; 2: 1-9. — https://antybiotyki.edu.pl/wp-content/uploads/2020/02/Biuletyn-NPOA-_2_2019.pdf
- See also: Food and Drug Administration Orbactiv — https://www.accessdata.fda.gov/drugsatfda_docs/label/2016/206334s003lbl.pdf
- See also: European Medicines Agency Orbactiv. — https://www.ema.europa.eu/en/medicines/human/EPAR/orbactiv